CLINICAL TRIAL: NCT04338984
Title: Combined Erector Muscle Spinae Plane Block and General Anaesthesia Versus General Anaesthesia Alone - Effect on Perioperative Opioid Consumption in Open Heart Surgery
Brief Title: Nociception-directed Erector Muscle Spinae Plane Block in Open Heart Surgery
Acronym: NESP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu (Other)
Responsible Party: Principal Investigator, Balan Ion Cosmin, Consultant in Cardiovascular Anaesthesia and ICM, Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18750
Record Dates: First submitted 2020-04-02; First posted 2020-04-08 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Regional Anesthesia; Heart Surgery
Keywords: erector spinae plane block; fast-track; rehabilitation; opioid
MeSH Terms: interventions — Anesthetics, General; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia alone (AG) (Active Comparator): Opioid based analgesia:
  Fentanyl 5 mcg/kg is standard dose at induction. Further dosing is steered according to NOL index and ancillaries such as heart rate and mean arterial blood pressure (± 20% of preoperative baseline).
  Postoperatively, analgesia comprises on-demand morphine and regularly dosed paracetamol.
  Interventions: Drug: General anesthetic
- Erector Spinae Plane Block and General Anaesthesia (ESPAG) (Experimental): Bilateral single shot erector spinae plane block with Ropivacaine 0.5% (total dose 3mg/kg) and Dexamethasone 8mg per every 20ml Ropivacaine 0.5% is performed before induction of general anaesthesia. A minimum 30 minutes interval is allowed before skin incision.
  Fentanyl 5 mcg/kg is standard dose at induction; rescue dosing is steered according to NOL index and ancillaries such as heart rate and mean arterial blood pressure (± 20% of preoperative baseline).
  Postoperatively, analgesia comprises on-demand morphine and regularly dosed paracetamol.
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution

INTERVENTIONS:
Drug: General anesthetic — Fentanyl is administered at induction - standard dose 5 mcg/kg. Further dosing is based on a multiderivative assessment of nociception (NOL index) and ancillaries such as heart rate and mean arterial blood pressure.
  Other Names: Fentanyl based general anaesthesia
  Arms: General anesthesia alone (AG)
Drug: Ropivacaine 0.5% Injectable Solution — Bilateral single shot erector spinae plane block is performed before induction of general anaesthesia.
  Ropivacaine 0.5% total dose 3mg/kg with Dexamethasone 8mg/20 ml Ropivacaine 0.5%.
  Other Names: Erector Spinae Plane Block
  Arms: Erector Spinae Plane Block and General Anaesthesia (ESPAG)

SUMMARY:
With the advent of ultrasound (US) guidance, use of regional anaesthesia (RA) is poised to grow and evolve. Recently, cardiac surgery has benefited from newer US guided interfascial techniques as they promise to fulfil all the prerequisites of an enhanced recovery after surgery (ERAS) strategy(1,2).

The erector spinae plane (ESP) block represents such an alternative(3). Speed and ease of performance are paramount to encourage spread of its use. Hence, the scope of this trial is to investigate the effects on perioperative opioid consumption and several other secondary outcomes of a minimalist approach encompassing a bilateral single shot ESP block when applied as an adjunct to general anaesthesia.

DETAILED DESCRIPTION:
DETAILED DESCRIPTION OF STUDY

A. Ethics

Local Ethics Committee approval and Informed Consent from patient or next-of-kin are obtained prior to study enrolment.

B. Study enrolment

Eighty adult patients scheduled for elective open cardiac surgery under general anaesthesia (GA) are randomly allocated to receive either GA plus ESP block (ESP group, n = 40) or GA alone (control group, n = 40).

C. Methods - Preinduction

1. Premedication with intramuscular morphine 0.1mg/kg 30 minutes before induction.
2. 16-G peripheral intravenous cannula and radial artery catheter.
3. Five-lead ECG, pulse oximetry, non-invasive and invasive blood pressure monitoring.
4. Analgesia monitor - the NoL index (PMD200TM, Medasense) finger probe will be connected to the index finger of the non-cannulated hand.
5. Surgical antibiotic prophylaxis (Cefuroxime 1.5g)
6. Stress ulcer prophylaxis (omeprazole 40 mg)

D. Methods - ESP block (intervention group only)

Before induction, patients in the intervention group are placed in sitting position under the close supervision of the attending nurse anaesthetist. After skin asepsis with chlorhexidine 2%, a high-frequency linear ultrasound probe is positioned parasagittally, 2-3 cm from midline, bilaterally, at the level of the T5 transverse process. A 25-G echogenic block needle is inserted at 20⁰-30⁰ in a caudal-to-cephalad direction until the tip of the needle reaches the interfascial plane between the erector spinae muscle and the inter-transverse ligaments. Correct hydrodissection at T5 level is first certified using normal saline. Subsequently, ropivacaine 0.5% with dexamethasone 8mg/20ml is used and maximum spread is attained by slowly advancing the needle as the interfascial plane splits up ahead. A maximum dose of 3mg/kg ropivacaine is used, corresponding to 1.5 mg/kg per side (e.g., 20 ml ropivacaine 0.5% / side for a 70kg adult). Supine position is resumed after completion of block.

E. Methods - General anaesthesia

1. End tidal CO2 (ETCO2).
2. Bispectral index (BIS) monitoring of hypnotic depth (target 40-60).
3. The nociception monitor (PMD200TM, Medasense) is started after induction of general anaesthesia; a calibration period of 1-2 minutes is usually required.
4. CVP insertion into the right internal jugular vein under ultrasound guidance. Any other hemodynamic monitor deemed useful is left at the discretion of the treating anaesthetist.
5. Urinary catheter, rectal temperature probe placement.
6. Intubating conditions

   6.1. Propofol 1-1.5 mg/kg or Etomidate 0.2-0.3 mg/kg.

   6.2. Fentanyl 5 mcg/kg.

   6.3. Atracurium 0.5 mg/kg.
7. Maintenance of anaesthesia

7.1. Sevoflurane in O2 during periods of preserved pulmonary blood flow and mechanical ventilation according to BIS (see target above).

7.2. Propofol infusion according to BIS (see target above) during periods of extracorporeal support.

7.3. Atracurium 0.2-0.3 mg/kg/h for adequate neuromuscular blockade.

7.4. Management of analgesia divides in:

7.4.1. Analgesia support

7.4.1.1. ESP block in the intervention group only:

• Theoretical duration of ESP block with surgical intensity is 4-6 hours.

7.4.1.2. Fentanyl (both study groups):

* Analgesia monitoring (see below) provides feedback to its administration.
* Administration follows a combination of continuous infusion and bolus dosing according to our local protocol:

  * Fentanyl 1.5 mg/50ml (30 mcg/ml).
  * Bolus dose (ml): Weight/20, which is equivalent to 1.5 mcg/kg.
  * Infusion rate (ml/hour): Weight/10, which is equivalent to 3 mcg/kg/h.
  * Last infusion rate before large vessel cannulation is maintained throughout the bypass period.

7.4.1.3. Paracetamol (both study groups):

• Administration of 2 grams following induction of general anaesthesia.

7.4.2. Analgesia monitoring

7.4.2.1. NoL index provides a multiderivative assessment of nociception before large vessel cannulation; depending on the spontaneous cardiac rhythm, it may be expected to continue reflecting nociception even after completion of extracorporeal circulation.

* Optimal analgesia is defined as a NoL index of 10-25.
* Allow periods of fluctuation of less than 1 minute.
* After sternotomy, allow a maximum fluctuation interval of 3 minutes before vital data are gathered.
* In the ESP group, if NOL target is attained, stop fentanyl administration.

7.4.2.2. Ancillaries such as mean arterial blood pressure (MAP) and heart rate (HR) provide complementary decision loops: targets are within ± 20% of preoperative baseline.

* During CBP they provide the only feedback on adequacy of analgesia, although highly unspecific.
* May be used at any time to complement the NoL index.

F. Methods - Postoperatively

1. Criteria to be met before extubation:

   1.1. Normothermia (T◦ ≥ 36◦C).

   1.2. No clinical bleeding.

   1.3. Wakefulness and RASS [-1;1].

   1.4. Hemodynamic stability with minimal vasoactive support (dobutamine < 5 µg/kg/min and norepinephrine < 100 ng/kg/min):

   1.4.1. MAP ≥ 60 mmHg

   1.4.2. Lactate ≤ 2 mmol/L

   1.4.3. Preserved flow (CI ≥ 2.2L/min/m2) assessed by:

   1.4.3.1. TTE any time after ICU admission

   1.4.3.2. TOE only before extubation, regardless of patient location

   1.5. Respiratory:

   1.5.1. Adequate gas exchange:

   1.5.1.1. Normocarbia.

   1.5.1.2. PaO2/FiO2 ≥ 250.

   1.5.2. Adequate effort:

   1.5.2.1. Tidal volume ≥ 5 ml/kg.

   1.5.2.2. Negative inspiratory force ≤ -20 cmH2O.

   1.5.3. Adequate airway reflex to handle secretions.
2. Management of analgesia divides in:

2.1. Analgesia support:

2.1.1. Paracetamol 1g iv 6 hourly is standard in both groups.

2.1.2. Morphine bolus doses of 0.03 mg/kg in combination with continuous iv morphine 0.03 mg/kg/h as elicited by nociception monitoring (see below).

2.2. Analgesia monitoring

2.2.1. The visual analogue scale (VAS) is used to provide feedback on adequacy of analgesia.

2.2.2. If VAS > 3, then provision of a combination of paracetamol and morphine is warranted (see above).

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent.
2. Elective heart surgery with sternotomy and bypass.
3. Hemodynamic stability prior to induction (no chest pain, SAP > 100 mmHg, MAP ≥ 60 mmHg, 50 < HR < 100 bpm).
4. Sinus rhythm.

Exclusion Criteria:

1. Known allergy to any of the medications used in the study.
2. BMI > 35.
3. Patient refusal to participate in the study.
4. Coagulopathy (INR > 1.5, APTT > 45, Fibrinogen < 150 mg/dl).
5. Non-elective/emergent and/or redo surgery.
6. ASA ≥ 4.
7. Any preoperative hemodynamic support (mechanical or pharmaceutical).
8. Severe LV dysfunction (LVEF ≤ 30%).
9. Severe RV dysfunction or PHT (RVFAC ≤ 25%).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Intraoperative fentanyl consumption (µg/kg/h) | during intraoperative period
  Goal directed monitoring of nociception with NOL index PMD200 (+/- variation of mean arterial blood pressure and heart rate)

SECONDARY OUTCOMES:
Fentanyl (µg/kg/h) consumption | until large vessel cannulation
  Goal directed monitoring of nociception with NOL index PMD200
Morphine consumption (mg/kg) | 24 hours and 48 hours after surgery
  Postoperative opioid administration
Quality of postoperative analgesia | 6 hours, 12 hours, 24 hours and 48 hours after extubation/ICU admission and 1 hour after drain removal
  Assessment - visual analog scale (VAS) (minimum of 0, maximum of 10)
Time to extubation | up to 24 hours after surgery
  Following ICU admission, the time it takes to extubate the patient safely
Norepinephrine dose (mcg/kg/h) | intraoperative, 6 hours and 12 hours after surgery
  Cumulative dose of Norepinephrine
Time to catecholamine - free state | up to 96 hours after surgery
  Following ICU admission, the time it takes to stop all catecholamines.
Rate of postoperative pneumonia | up to two weeks
  Postoperative incidence
Rate of atrial fibrillation | 48 hours after ICU admission
  Postoperative incidence
Time to first out of bed | up to 72 hours after surgery
Rate of nausea and vomiting (PONV) | 24 hours after ICU admission
Rate of delirium | 7 days after surgery
Time to removal of drain | up to 72 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Serban Ion Bubenek Turconi, Professor, Study Director — Prof. Dr. C.C. Iliescu Institute for Emergency Cardiovascular Diseases; Dana Tomescu, Professor, Study Director — Fundeni Clinical Institute
Locations (1):
- Prof Dr CC Iliescu Institute for Emergency Cardiovascular Diseases, Bucharest, Romania

REFERENCES:
- [Background] Smith LM, Barrington MJ; St Vincent's Hospital, Melbourne. Ultrasound-guided blocks for cardiovascular surgery: which block for which patient? Curr Opin Anaesthesiol. 2020 Feb;33(1):64-70. doi: 10.1097/ACO.0000000000000818. PMID 31833864
- [Background] Kelava M, Alfirevic A, Bustamante S, Hargrave J, Marciniak D. Regional Anesthesia in Cardiac Surgery: An Overview of Fascial Plane Chest Wall Blocks. Anesth Analg. 2020 Jul;131(1):127-135. doi: 10.1213/ANE.0000000000004682. PMID 32032103
- [Background] Macaire P, Ho N, Nguyen T, Nguyen B, Vu V, Quach C, Roques V, Capdevila X. Ultrasound-Guided Continuous Thoracic Erector Spinae Plane Block Within an Enhanced Recovery Program Is Associated with Decreased Opioid Consumption and Improved Patient Postoperative Rehabilitation After Open Cardiac Surgery-A Patient-Matched, Controlled Before-and-After Study. J Cardiothorac Vasc Anesth. 2019 Jun;33(6):1659-1667. doi: 10.1053/j.jvca.2018.11.021. Epub 2018 Nov 19. PMID 30665850